CLINICAL TRIAL: NCT05531266
Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cells as First-line Treatment for Patients With Acute Graft Versus Host Disease
Brief Title: Umbilical Cord Mesenchymal Stem Cells as First-line Treatment for Patients With Acute Graft Versus Host Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220831
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: aGVHD
Keywords: aGVHD; Umbilical Cord Mesenchymal Stem Cell
MeSH Terms: interventions — Glucocorticoids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hUC-MSCs combined with glucocorticoids group. (Experimental): 91 patients will be involved in this group
  Interventions: Other: hUC-MSCs
- glucocorticoids group (Active Comparator): 91 patients will be involved in this group
  Interventions: Other: glucocorticoids

INTERVENTIONS:
Other: hUC-MSCs — Participants will be treated with hUC-MSCs at a dose of 1×10^6 /kilogram (kg) actual body weight at Screening for twice per week in 1-2 weeks and once a week in 3-4 weeks after being rolled into this study. At the same time, patients will be treated with glucocorticoids according to patients' condition.
  Arms: hUC-MSCs combined with glucocorticoids group.
Other: glucocorticoids — Participants were treated with glucocorticoids only.
  Arms: glucocorticoids group

SUMMARY:
Allogenic haemopoietic stem cell transplantation (allo-HSCT) is the effective treatment for many hematologic malignancies and some non-malignant diseases. In recent years, with the rapid improvement of economy and medical level, the number of cases of hematopoietic stem cell transplantation (HSCT) develops rapidly in China. In 2019, 12,323 cases of HSCT were completed in China, with allo-HSCT accounting for 9600 cases of which.

However, Graft versus host disease (GVHD) is one of the most common and serious complications after Allo-HSCT. The incidence of acute GVHD (aGVHD) is as high as 40%-60% in HLA-matched sibling transplantation, and the incidence is even higher in haplo-hematopoietic stem cell transplantation(haplo-HSCT) and unrelated donor transplantation. By Glucksberg grading standard, the 5-year survival rates of grade III and IV aGVHD are 25% and 5% respectively, indicating severe GVHD directly affects the survival of Allo-HSCT patients.

The first-line treatment for aGVHD is still glucocorticoid, while the effective rate is only 30%-50%. Moreover, due to immunosuppression and increasing risk of infection, the efficacy of second-line treatments including polyclonal antibodies, monoclonal antibodies, immunosuppressants, immunotoxins, chemotherapy drugs, and light therapy for steroid resistant aGVHD is also poor, with the overall survival rate of 5%-30%.

Mesenchymal stem cells (MSCs) are multipotent cells, which can promote engraftment and hematopoietic reconstruction by secreting a variety of hematopoietic promoting factors, expressing adhesion molecules supporting hematopoietic stem cells, guiding homing of hematopoietic stem cells and providing hematopoietic microenvironment. At the same time, MSCs can modulate immune responses by affecting the proliferation of T cells and the migration of T cells and DC, inducing the expansion of Treg cells, inhibiting the secretion of antibodies by B lymphocytes, and regulating the secretion of soluble factors such as NO and IDO. As a result of these characteristics and the poor immunogenicity, MSCs are a promising alternative treatment for GVHD.

Currently, UK and EU guidelines has recommended MSC as a third-line treatment for grade 2-4 acute GVHD, and the safety and efficacy of umbilical cord derived MSCs in the prevention and treatment of GVHD has also been reported by several transplantation centers in China.However, MSCs have not been used for first-line treatment of aGVHD. Therefore, the investigators designed this study to evaluate the safety and efficacy of UC-derived MSCs as the first line treatment in patients with aGVHD.

DETAILED DESCRIPTION:
This prospective, randomized and controlled study is to investigate the efficacy and safety of Umbilical Cord Mesenchymal Stem Cells as First-line Treatment for Patients With Acute Graft Versus Host Disease. Investigators will recruit 182 patients with acute leukemia, with 91 of them entering the hUC-MSCs combined with glucocorticoids group. and receiving hUC-MSCs at a dose of 1×10^6 /kilogram (kg) actual body weight at Screening for twice per week in 1-2 weeks and once a week in 3-4 weeks after being rolled into this study, with the glucocorticoid given at the same time. while the other 91 entering the glucocorticoids group receiving glucocorticoids only. Then primary outcomes including the ORR at day 180 post initiation of therapy, as well the secondary outcomes including cumulative relapse incidence、cumulative incidence of chronic GVHD 、cumulative Incidence of infectious complications and cumulative Incidence of lymphoproliferative disease will be measured during 180 days after the intervention being finished.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has undergone an allogeneic haematopoietic stem cell transplantation (HSCT) and developed acute graft versus host disease (aGVHD)
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* serum creatinine less than twice the upper limit of normal or creatinine clearance greater 50 ml/min within 28 days.
* Patients had recovered from previous treatments
* Signing written informed consent and agreeing with taking designated umbilical cord blood

Exclusion Criteria:

* Patients had severe allergy history
* Patients with unstable angina or whose cardiac function grading III-IV.
* Patients with chronic respiratory disease requiring continuous oxygen supplement
* Patients with active hepatitis B or active hepatitis C or AIDS infection
* Patients with Uncontrolled viral or bacterial infections
* Patients with severe psychiatric or physical illness that would limit compliance with study requirements
* Patients who received any other investigational study or treatment within 30 days
* Secondary malignancy
* Allergic to blood products
* Other causes which are not suitable for the trial in investigator's consideration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Day 28 Post Initiation of Therapy | 28 days
  ORR was defined as the percentage of participants who had achieved overall response. Overall response was defined as complete response (CR) plus partial response (PR) according to aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ.

SECONDARY OUTCOMES:
Cumulative relapse incidence | 180 days
  Defined as the cumulative incidence of relapse after the day of transplantation.
cumulative incidence of chronic GVHD at one year | 180 days
  chronic graft versus host disease will be diagnosed and graded by National Institute of Health Consensus (NIH Consensus).
Cumulative Incidence of Infectious Complications | 180 days
  Defined as cumulative incidence of viral, fungal and bacterial infections.
Cumulative Incidence of lymphoproliferative disease | 180 days
  Defined as the cumulative incidence of lymphoproliferative disease after the day of transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China